CLINICAL TRIAL: NCT01734733
Title: A Phase I/IIa, Open-label Investigation of the Safety and Clinical Effects of NTCELL [Immunoprotected (Alginate-Encapsulated) Porcine Choroid Plexus Cells for Xenotransplantation] in Patients With Parkinson's Disease
Brief Title: Open-label Investigation of the Safety and Clinical Effects of NTCELL in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Living Cell Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCT/PD-012
Record Dates: First submitted 2012-11-18; First posted 2012-11-28 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Xenotransplantation; choroid plexus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NTCELL (Experimental): NTCELL 40 microcapsules (+/- 20%)
  The NTCELL microcapsules are drawn up into a catheter system and introduced intracranially by stereotactic insertion into the brain under guidance by neuroimaging.
  Interventions: Other: NTCELL

INTERVENTIONS:
Other: NTCELL

SUMMARY:
To assess the safety of xenotransplantation of NTCELL [immunoprotected (alginate-encapsulated) choroid plexus cells] in patients with Parkinson's disease, assessed over the duration of the study, by monitoring the occurrence of adverse events and serious adverse events, including clinical and laboratory evidence of xenogeneic infection in transplant recipients and their partners/close contacts. Subsequent safety follow-up will include lifelong monitoring for clinical and laboratory evidence of xenogeneic infection.

To assess the clinical effects of NTCELL [immunoprotected (alginate-encapsulated) choroid plexus cells] in patients with Parkinson's disease. This will be quantified by testing the secondary endpoints of the trial as described below (see Endpoints/Outcome Measures).

DETAILED DESCRIPTION:
Parkinson's disease is characterized by widespread neural degeneration, particularly in the substantia nigra and its projections to the basal ganglia. Current therapy for Parkinson's disease is purely symptomatic. There is a pressing need for a treatment that reverses or slows the degeneration of the nigrostriatal pathway.

Numerous transplant-based therapies have attempted to support, repair or replace the degenerating nigrostriatal neurons. These have included the transplantation of foetal and other neuronal stem cells, gene transfers, and the implantation of devices releasing neural growth factors. All these have been shown to have some effectiveness in animal models, but have been generally disappointing in human studies.

Intracranial choroid plexus cell transplantation has the potential to deliver biological neural agents for the treatment of Parkinson's disease which cannot be achieved by conventional treatment. The overall aim of delivering neural proteins and compounds over many months to the basal ganglia of the brain is to enhance neural repair currently not possible with antiparkinsonian medication or deep brain stimulation (DBS).

As animal-derived tissues have to be protected from immune rejection when transplanted into humans, transplants are usually accompanied by immunosuppressive therapy. However, porcine choroid plexus cells are preferably implanted without the use of immunosuppressive drugs which cause significant morbidity. To protect them from immune rejection, the cells can be encapsulated in alginate microcapsules which permit the inward passage of nutrients and the outward passage of biologic neural proteins and compounds normally secreted by choroid plexus cells. Alginate-encapsulated porcine choroid plexus cells implanted into the brain without immunosuppressive drugs have survived rejection for many months in animal studies.

NTCELL comprises neonatal porcine choroid plexus cells encapsulated in alginate microcapsules. NTCELL has been safely implanted in rats, and non-human primates. Following NTCELL implants, animals with chemically-induced Parkinson's-like lesions showed improvement of functional neurological motor abnormalities that was associated with histologic changes consistent with amelioration of the lesion.

The initial dose for intracranial implantation of the current NTCELL preparation for the treatment of Parkinson's disease in humans is based on the effective dose in a non-human primate (rhesus monkey) model.

Parkinson's disease patients will be followed up for 26 weeks after receiving an implantation of NTCELL administered into the putamen of the corpus striatum on the side contralateral to the greatest clinical deficit.

Based upon the data obtained during the 26-week follow-up period a decision will be made as to whether the patient will receive:

* an implantation of a second dose of NTCELL
* unilateral DBS
* bilateral DBS
* no further intervention

The data will be reviewed by the investigators and the Data Safety Monitoring Board (DSMB), the data will consist of clinical outcomes and clinimetric data, an MRI scan, PET scanning, and adverse events.

Patients will be followed up for a further 48 weeks if there is no further intervention, however if it is decided that either DBS or implantation of a second dose of NTCELL occurs then the frequency of follow-up will be the subject of a protocol amendment.

ELIGIBILITY:
Inclusion Criteria:

To be assessed at the Week -10 to -4 Visit

* Adults (males or females) in the age range 40 to 70 years
* Diagnosis of Parkinson's disease (minimum duration of 5 years) in accordance with the London Brain Bank criteria
* Patients diagnosed with idiopathic Parkinson's disease
* Stable medication for Parkinson's for at least 1 month
* Patients with advanced and fluctuating Parkinson's disease who have met the criteria for DBS and who have been accepted for DBS at Auckland City Hospital. These criteria include exhaustion of available medication treatments for Parkinson's disease, normal brain MRI, intact cognitive, psychological and psychiatric function, appropriate carer support, and competence and willingness to consent to the placement of deep brain probes
* If female, no childbearing capability (those who are more than 2 years postmenopausal or have undergone voluntary sterilisation can be considered for enrolment)
* Provision of written informed consent. Patients will be required to agree to comply with all tests and visits specified in the protocol, and they (and their partners/close contacts) will also be required to consent to long-term microbiological monitoring, which is an integral part of the study.

Exclusion Criteria:

To be assessed at the Week -10 to -4 Visit

Note: the criteria for acceptance for DBS would exclude patients with comorbidities that normally would exclude them from similar studies, including uncontrolled depression, dementia, focal neurological deficits, or secondary parkinsonism. Specific exclusion criteria in this category are:

* Any history of central nervous system infection
* Significant dementia as determined by neuropsychological assessment
* Focal neurological defects
* Evidence of significant medical or psychiatric disorders
* Secondary parkinsonism
* Severe autonomic symptoms
* Atypical Parkinson's disease
* History of substance abuse
* Body mass index (BMI) ≥30 kg/m2 or ≤20 kg/m2
* Serious comorbid conditions that are likely to affect participation in the study, including:

  * Previous coronary heart disease manifesting as non-ST elevation myocardial infarction (NSTEMI), Q-wave infarction or unstable angina; coronary artery bypass graft (CABG); or percutaneous angioplasty
  * Previous cerebrovascular disease manifesting as transient ischaemic attacks (TIAs) or stroke
  * Peripheral vascular disease with foot ulcer and/or previous amputation
  * History of New York Heart Association (NYHA) class II, III or IV congestive heart failure (CHF) and/or chronic atrial fibrillation
  * Chronic obstructive pulmonary disease (COPD) or asthma with previous hospitalisation for decompensation; a requirement for mechanical ventilation at any stage; or long-term treatment with oral corticosteroids
  * Liver disease with abnormal liver function tests defined as serum bilirubin ≥20 µmol/L, and/or ALT ≥100 U/L, and/or GGT ≥100 U/L, and/or albumin < 35 g/L
  * Haematological disorders, including haemoglobin ≤110 g/L or platelet count < 80 x 109/L
  * Kidney disease, defined as serum creatinine > 130 μmol/L in men and > 110 μmol/L in women and/or haematuria and/or active urinary sediment or casts
  * Peptic ulcer disease and/or history of previous gastrointestinal bleeding
  * Malignancy other than basal cell carcinoma
  * History of epilepsy
  * Untreated hypothyroidism
  * Known adrenal insufficiency

Other exclusion criteria:

* Past history of brain surgery for Parkinson's disease
* Poor candidate for any surgery
* HIV antibody and/or risk factors for HIV infection
* Positive hepatitis C antibody, positive hepatitis B surface antigen, and hepatitis B core antibody
* Current administration of immunosuppressive medications (e.g. cyclosporin, tacrolimus, sirolimus, mycophenolate mofetil, muromonab-CD3, daclizumab, basiliximab, antithymocyte globulin, interferons) for other disease conditions
* Inability to travel on aeroplane to Vancouver (for PET scan)
* Any other condition that, in the opinion of the Investigator, may interfere with adherence to the study protocol.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-07-12 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2020-06-04 (Actual)

PRIMARY OUTCOMES:
the safety of xenotransplantation of NTCELL | 26 weeks
  measured by the incidence of adverse events, clinical laboratory tests (including xenogeneic viral analysis), physical examination, review by infectious disease physician

SECONDARY OUTCOMES:
Brain metabolism as demonstrated on PET with [18F]-fluorodopa measured at 26 weeks post-implant 1 compared with baseline | 26 weeks
Brain metabolism as demonstrated on PET with [11C]-tetrabenazine measured at 26 weeks post-implant 1 compared with baseline | 26 weeks
Scores measured by the Unified Parkinson's Disease Rating Scale (UPDRS Parts I, II, III, IV - Parts II and III will be performed in the 'off' and 'on' state) over 26 weeks post-implant 1 compared with the baseline scores | 26 weeks
Modified Hoehn and Yahr stages over 26 weeks post-implant 1 compared with the baseline stages | 26 weeks
Scores measured by the Unified Dyskinesia Rating Scale (UDysRS Parts I, II, III, IV - Parts III and IV will be performed in the 'off' and 'on' state) over 26 weeks post-implant 1 compared with the baseline scores | 26 weeks
Times for hand-arm movement between 2 points (tapping test) in accordance with the CAPSIT-PD protocol (Defer et al. 1999) over 26 weeks post-implant 1 compared with the baseline times | 26 weeks
Scores measured by the modified walking test in accordance with the CAPSIT-PD protocol (Defer et al. 1999) (walking 4.5m back and forth instead of 7m back and forth) over 26 weeks post-implant 1 compared with the baseline scores | 26 weeks
Scores measured by the Parkinson's Disease Questionnaire (PDQ-39) over 26 weeks post-implant 1 compared with the baseline scores | 26 weeks
Scores measured by neuropsychological tests at 26 weeks post-implant 1 compared with the baseline scores | 26 weeks
  TESTS USED
  * National Adult Reading Test
  * Speed and Capacity of Language Processing Test
  * Boston Naming Test
  * Trail Making Test A
  * Trail Making Test B
  * WMS IV Logical Memory I
  * WMS IV Logical Memory II
  * RAVLT List Learning
  * RAVLT Short Delay Recall
  * RAVLT Long Delay Recall
  * Rey Complex Figure Copy
  * Rey Complex Figure Delayed Recall
  * WAIS IV Digit Span
  * WAIS IV Matrix Reasoning
  * WAIS IV Symbol Search
  * WAIS IV Coding
  * DKEFS Word Fluency
  * DKEFS Category Fluency
  * DKEFS Category Switching
  * DKEFS Colour Naming
  * DKEFS Word Reading
  * DKEFS Inhibition
  * DKEFS Inhibition/switching
  * Mini Mental State Examination
  * Montreal Cognitive Assessment
  * HADS Anxiety
  * HADS Depression
Psychiatric assessment at 26 weeks post-implant 1 compared with the baseline psychiatric assessment | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Barry Snow, MBChB, Principal Investigator — Auckland City Hospital
Locations (1):
- Auckland City Hospital, Auckland, New Zealand